CLINICAL TRIAL: NCT00216346
Title: A Phase 3 Multicenter, Randomized, Controlled, Clinical Trial to Assess the Safety and Efficacy of Injectable Paromomycin in Patients With Visceral Leishmaniasis
Brief Title: Safety and Efficacy Study of Paromomycin to Treat Visceral Leishmaniasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: World Health Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VLPM01
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Visceral Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — Paromomycin; Amphotericin B

INTERVENTIONS:
Drug: Paromomycin sulfate
Drug: Amphotericin B

SUMMARY:
Symptomatic Visceral Leishmaniasis(VL)is fatal; Due to the increasing resistance to standard therapy with antimonials, there is a need for new safe, efficacious, low-cost therapies for the treatment of VL. Paromomycin is an off-patent aminoglycoside antibiotic with anti-leishmaniasis activity. This study will test the safety and efficacy of paromomycin in the treatment of patients with VL in India.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5-55 years (inclusive) of either gender.
* Newly diagnosed VL or VL treatment failure confirmed by spleen or bone marrow aspirate.
* Clinical signs and symptoms compatible with VL: fever of over two weeks duration and splenomegaly.
* Biochemical and haematological test values as follows:

  * Haemoglobin > 5.0g/100mL
  * White blood cell count > 1 x109/L
  * Platelet count > 50 x 109/L
  * AST, ALT and alkaline phosphatase < 3 times upper normal limit
  * Prothrombin time < 5 seconds above control
  * Serum creatinine levels within normal limits
  * Serum potassium levels within normal limits
* HIV negative

Exclusion Criteria:

* A history of intercurrent or concurrent diseases (e.g. chronic alcohol consumption or drug addiction; renal, hepatic, cardiovascular or central nervous system disease; diabetes; tuberculosis or other infectious or major psychiatric diseases) that may introduce variables affecting the outcome of the study.
* Any condition which the investigator thinks may prevent the patient from completing the study therapy and subsequent follow-up.
* An abnormal baseline audiogram (presentation with 75 dB or higher at 8KHz or below) and/or a history of significant vestibular or auditory dysfunction.
* Proteinuria (> 2+).
* A history of allergy or hypersensitivity to aminoglycosides.
* A history of major surgery within the last two weeks.
* Pregnancy or lactation. [Note: women of childbearing age must use an adequate form of contraception (documented) or agree to a period of sexual abstinence during the treatment phase of the study.]
* Previous treatment for VL within two weeks of enrolment into the study.
* Prior treatment failures with paromomycin or amphotericin B.

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 667
Dates: Start 2003-06; Study Completion 2004-11

PRIMARY OUTCOMES:
(1) To compare the safety of injectable paromomycin to amphotericin B when administered in the proposed dosage regimens.
(2) To compare the efficacy of injectable paromomycin to amphotericin B with regards to final cure rates.

SECONDARY OUTCOMES:
- Characterization of the pharmacokinetics of injectable paromomycin in adults and children with VL
- Comparison of initial cure rates for the two regimens
- Comparison of clinical improvement rates for the two regimens

CONTACTS AND LOCATIONS:
Overall Officials: Prof S. Sundar, Principal Investigator — Kala-azar Research Centre; Prof T.K. Jha, Principal Investigator — Kalazar Research Centre; Prof C.P. Thakur, Principal Investigator — Kalazar Research Centre; Dr. S.K. Bhattacharya, Principal Investigator — Rajendra Memorial Research Institute of Medical Sciences (ICMR)
Locations (4):
- India (4):
  - Rajendra Memorial Research Institute of Medical Sciences (ICMR), Agam Kuan, Patna, Bihar
  - Kalazar Research Centre, Brahmpura, Muzaffarpur, Bihar
  - Kalazar Research Centre, Patna, Bihar
  - Kala-azar Medical Research Centre, Rambagh Road Muzaffarpur, Bihar

REFERENCES:
- [Derived] Sundar S, Jha TK, Thakur CP, Sinha PK, Bhattacharya SK. Injectable paromomycin for Visceral leishmaniasis in India. N Engl J Med. 2007 Jun 21;356(25):2571-81. doi: 10.1056/NEJMoa066536. PMID 17582067